CLINICAL TRIAL: NCT02691598
Title: Dexmedetomidine Hydrochloride in the Prevention of Organ Failure Following
Brief Title: Dexmedetomidine Hydrochloride in the Prevention of Organ Failure Following Severe Acute Pancreatitis
Acronym: DHPOFFSAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Nanjing University School of Medicine (Other)
Responsible Party: Principal Investigator, Weiqin Li, Dr., Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: DHPOFFSAP1
Record Dates: First submitted 2016-02-14; First posted 2016-02-25 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Pancreatitis, Acute Necrotizing
MeSH Terms: conditions — Pancreatitis, Acute Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Dexmedetomidine Hydrochloride 4ug/ml；0.05ml/kg.h infusion for 24hours
  Interventions: Drug: Infusion
- Group B (Placebo Comparator): Normal Saline 0.05ml/kg.h infusion for 24hours
  Interventions: Drug: Infusion

INTERVENTIONS:
Drug: Infusion — Dexmedetomidine Hydrochloride or normal saline 4ug/ml；0.05ml/kg.h infusion for 24hours
  Other Names: yan suan you meituo mi ding zhu she ye

SUMMARY:
Cytokines such as such as TNF-a, IL-1, IL-6 correlate with the severity of pancreatitis.Neuroendocrine pathways, such as the sympathetic nervous system or parasympathetic nervous system, in turn, have some impact on the immune systems, through a-2 adrenoreceptor stimulation or the cholinergic anti-inflammatory pathway. The investigators aim to use Dexmedetomidine Hydrochloride to decrease the activity of sympathetic nervous system, thus relieve inflammation response.

DETAILED DESCRIPTION:
Infected pancreatic necrosis (IPN) and multiple organ dysfunction syndrome (MODS) are major complications of acute pancreatitis which determine disease severity and outcome.It is concluded that systemic inflammation in SAP characterized by the endocrine release of different cytokines, such as TNF-a, IL-1, IL-6 and many others. These cytokines correlate with the severity of pancreatitis.

Neuroendocrine pathways, such as the sympathetic nervous system or parasympathetic nervous system, in turn, have some impact on the immune systems, through a-2 adrenoreceptor stimulation or the cholinergic anti-inflammatory pathway. Dexmedetomidine Hydrochloride is a high selected a-2 adrenoreceptor agonists.Some studies have shown that Dexmedetomidine Hydrochloride could improve the outcome of sepsis patients and decrease the development of organ failure.

The investigators aim to use Dexmedetomidine Hydrochloride to decrease the activity of sympathetic nervous system,thus relieve inflammation response.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with severe acute pancreatitis within 48h
* APACHE II≥8
* Patients or the family agreed to receive the treatment, and signed the informed consents

Exclusion Criteria:

* Patients were allergy to the drug
* Patients were diagnosed with Arrhythmia
* Patients with artificial permanent pacemaker implantation

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 314 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-02 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of Organ failure | 30 days after Incidence of the disease

SECONDARY OUTCOMES:
Infected pancreatic necrosis | 30 days after Incidence of the disease

CONTACTS AND LOCATIONS:
Overall Officials: Weiqin Li, M.D., Study Director — Jinling Hospital, China
Locations (1):
- Department of SICU, Research Institute of General Surgery Jinling Hospital, Nanjing, Jiangsu, China, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Zhang L, Zhou J, Ke L, Nie Y, Tong Z, Li W, Li J. Role of heart rate variability in predicting the severity of severe acute pancreatitis. Dig Dis Sci. 2014 Oct;59(10):2557-64. doi: 10.1007/s10620-014-3192-5. Epub 2014 May 13. PMID 24821463